CLINICAL TRIAL: NCT03400761
Title: Does Body Composition Predict Running Time?
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Genton Graf Laurence, Assistant Professor, University Hospital, Geneva
Other Study IDs: 2017-01327
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Body Composition; Running Performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several studies performed in elite endurance athletes have shown that running performance may be determined by a low fat mass in the overall population.

The "Course de l'Escalade" occurs yearly during the first week-end of December. This race takes place in the city of Geneva. The distance of this race is 7.3 km for all men and elite women, and 4.8 km for non-elite women. During this race, measurement of body composition by biolelectrical impedance analyses (BIA) were performed in volunteer, between December 1999 and 2017.

Hypothesis :

We hypothesize that:

1. A low fat mass is associated with a slower running time, when adjusting for age, body weight, and habitual physical exercise.
2. An increase in fat mass over time increases running time over the years

Objectives :

1. To evaluate whether total and regional body composition is associated with running time at the "Course de l'Escalade".
2. To determine whether changes in body composition with progressive aging lead to changes in running time.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who underwent a measurement of body composition by tetrapolar bioelectrical impedance analyses (BIA) at the "Course de l'Escalade", a fun race occurring yearly in Geneva, between December 1999 and 2017.

Exclusion Criteria:

* Measurements of people <18 years at the time of BIA measurement.
* Measurements of people who did not perform or finish the race.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a historical cohort study of prospectively collected measurements of body composition performed by bioelectrical impedance analysis (BIA) at the "Course de l'Escalade", between 1999 and 2017. The "Course de l'Escalade" is a fun race occurring yearly in Geneva, between December 1999 and 2017. The distance of this race is 7.3 km for all men and elite women, and 4.8 km for non-elite women.
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Actual)
Dates: Start 1999-12-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Association between total and regional body composition and running time at the "Course de l'Escalade" | One day per year between 1999 and 2017 (i.e. the day of the "Course de l'escalade")
  Body composition measured by bioelectrical impedance analyses. Running time timed.

SECONDARY OUTCOMES:
Association between changes in body composition with progressive aging and changes in running time at the "Course de l'Escalade" | One day per year between 1999 and 2017 (i.e. the day of the "Course de l'escalade")
  Body composition measured by bioelectrical impedance analyses. Running time timed.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Genton, Pr. Dr. med, Principal Investigator — University Hospital, Geneva

REFERENCES:
- [Derived] Genton L, Mareschal J, Norman K, Karsegard VL, Delsoglio M, Pichard C, Graf C, Herrmann FR. Association of phase angle and running performance. Clin Nutr ESPEN. 2020 Jun;37:65-68. doi: 10.1016/j.clnesp.2020.03.020. Epub 2020 Apr 15. PMID 32359757